CLINICAL TRIAL: NCT02544178
Title: EPIBRAINRAD : Study of Neurological Complication After Radiotherapy for Glioblastoma High Grade
Brief Title: Study of Neurological Complication After Radiotherapy for High Grade Glioblastoma
Acronym: EPIBRAINRAD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sophie JACOB (Other Government)
Collaborators: Centre National de la Recherche Scientifique, France (Other)
Responsible Party: Sponsor-Investigator, Sophie JACOB, Dr, Institut de Radioprotection et de Surete Nucleaire
Organization: Institut de Radioprotection et de Surete Nucleaire (Other Government)
Other Study IDs: IRSN_02
Record Dates: First submitted 2015-07-20; First posted 2015-09-09 (Estimated); Last update posted 2016-09-22 (Estimated); Status verified 2016-09

CONDITIONS: Leukoencephalopathy
Keywords: radiotherapy; neurocognitive defect; leukoencephalopathy
MeSH Terms: conditions — Leukoencephalopathies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — * protéin S-100B, 8,12-iso-iPF2α-VI level, homocystéine
  * micro RNAs (brain-miR-112, brain-miR-161, hsa-let-7d-3p, hsa-miR-5010-3p, hsa-miR-26a-5p, hsamiR-1285-5p, hsa-miR-151a-3p, hsamiR-103a-3p, hsa-miR-107, hsa-miR-532-5p, hsa-miR-26b-5p, hsa-let-7f-5p, …).
  * microparticules
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- diagnostic procedure: neurocognitive tests before and after radiotherapy
  Interventions: Radiation: brain radiotherapy

INTERVENTIONS:
Radiation: brain radiotherapy — effect of cerebral radiotherapy on neurocognitive state

SUMMARY:
The survival time and the number of long time survivors after radiotherapy in brain cancer patients have increased for the last decades. Therefore the topic of late-delayed neurotoxic effects of this therapy gains more and more importance. Among these side effects, the main and most frequent one is the leukoencephalopathy, a diffused and progressive damage of the white matter characterized by myelin loss, loss of axons and vascular lesions. The incidence rate assessment, as well as the occurrence time, is based on retrospective studies with low numbers of patients, but seems to reach 30 to 50 % of the patients according to the follow-up. The risk seems to be increased during the first two years after the radiotherapy, but persists for decades.

To gain further insight in the radiation-induced leukoencephalopathy, the objective of this project is to study the onset and evolution of leukoencephalopathy in a 3-year prospective cohort of patients having undergone cerebral radiotherapy for glioma (stage 3-4), using specific cognitive tests, Magnetic Resonance Imagery (MRI) scans of the brain and predictive bio-markers of cognitive impairments.

DETAILED DESCRIPTION:
Context The survival time and the number of long time survivors after radiotherapy in brain cancer patients have increased for the last decades. Therefore the topic of late-delayed neurotoxic effects of this therapy gains more and more importance. Among these side effects, the main and most frequent one is the leukoencephalopathy, a diffused and progressive damage of the white matter characterized by myelin loss, loss of axons and vascular lesions. The incidence rate assessment, as well as the occurrence time, is based on retrospective studies with low numbers of patients, but seems to reach 30 to 50 % of the patients according to the follow-up. The risk seems to be increased during the first two years after the radiotherapy, but persists for decades.

No complete characterization of this cognitive impairment has been done yet due to crucial discrepancies in the neuropsychological assessments that were used (namely missing of pre-treatment assessment), in the follow-up of patients and in the applied treatment. However, based on previous studies, it can be said that the short term memory and the frontal functions are mainly affected and the quality of life is exceedingly impaired. Irradiation schemes, in particular high doses and large irradiated volume, have been identified as risk factors of leukoencephalopathy. However, in spite of modified protocols that tended to limit the risk, the remaining occurrence of the disease suggests a high dependency on individual risk factors, that are still poorly known and make the individual sensitivity to develop these secondary effects unpredictable. Other factors such as cardio-vascular factors, smoking, old age and combined radio-chemotherapy are linked to leukoencephalopathy as well, although only few of these associations were proved in large studies. Moreover, some specific bio-markers could complete clinical examinations to predict risk of cognitive impairment in these patients. Several biomarkers could be of interest:

The protein S-100B is a protein synthesized mainly by glial cells and cells of Schwann. It is an intracellular protein regulating the cytosolic availability of calcium. Its concentration is 30-100 times brought up in the cerebral tissue that in the other tissues. Its plasmatic half-life is a 1 hour, its elimination is renal. So, the protein S-100B is a marker of traumatic brain injury, certain neurodegenerative disorders and malignant gliomas. The dosage maybe so realized in serum and urines.

* Growing evidence implicates oxidative/nitrative damage in the pathogenesis of neurodegenerative disorders. Subsequent studies were undertaken showing that specific isoprostanes (iPs) levels are elevated in urine and blood of Alzheimer Disease patients and that these values correlate with memory impairments. This suggests that iPs are useful biomarkers in neurological diseases. Their levels could be measured in urine and plasma of patients.
* Homocysteine is a sulfur-containing amino acid, derived from the metabolism of methionine. Higher levels of homocysteine were associated with worse memory performance in a large group of older subjects. While homocysteine is not a diagnostic test, it may represent a modifiable risk factor for dementia.

Highlighting neuropsychological disorders including at an early stage requires a reliable and reproducible assessment of the patient's cognitive state. However, a comprehensive neuropsychological assessment takes several hours and a qualified staff, making it difficult to implement in the conventional patient monitoring. The use of a simple and fast tool to detect cognitive impairment would help to develop a systematic approach for screening these disorders. A detection computerized neuropsychological standardized test (Computerized Cognitive Speed Test - CSCT) assessing processing speed of information, attention and working memory has been validated in multiple sclerosis patients compared to healthy volunteers. CSCT quickly detects patients with cognitive impairment, who could be then tested with more complete tests. It can be conducted by people with no neuropsychology training and the testing time is less than 2 minutes.

This study will allow a better understanding of the impact of cognitive sequelae in patients treated for glioma with current standard treatments, including radiation. The validation of a new screening test, the CSCT, in this disease will eventually detect earlier these effects and possibly initiate treatment before lesions are too advanced. Feasibility of the implementation of the CSCT in "routine" practice for all patients treated with brain radiotherapy will be tested.

• Objectives and methodology To gain further insight in the radiation-induced leukoencephalopathy, the objective of this project is to study the onset and evolution of leukoencephalopathy in a 3-year prospective cohort of patients having undergone cerebral radiotherapy for glioma (stage 3-4), using specific cognitive tests, MRI scans of the brain and predictive bio-markers of cognitive impairments.

Primary objective:

- To constitute a prospective cohort of patients treated for glioma (stage 3-4) with radiotherapy in order to estimate the incidence rate and occurrence time of the leukoencephalopathy at the end of the follow-up (3 years after first inclusion).

Secondary objectives:

* To validate the CSCT- Computerised Speed Cognitive Test to detect early cognitive impairment in this patients population compared with complete cognitive tests
* Estimate precisely the dose received by the different anatomical parts of the brain
* To study the relation between the risk of leukoencephalopathy and the received dose to the brain
* To analyze the prognostic risk factors of leukoencephalopathy (either linked to radiation treatment or to patients' clinical conditions) among patients with glioma (stage 3-4)
* To propose and test some bio-markers as predictive factors of cognitive impairment
* To study the radiological changes on MRI associated with neurological abnormalities
* To build a biological collection for patients treated in the Pitié Salpêtrière Hospital

Patients with a diagnostic of glioma (stage 3-4) treated with radiotherapy in 2 hospitals (Hospital Pitié Salpêtrière, Paris and Institut Paul Strauss, Strasbourg) will be eligible for the study.

Taking into account that about 100 patients with glioma are treated every year in the Radiation Oncologic department of the Pitié Salpêtrière Hospital and 50 in the Paul Strauss Institute, the inclusion of 200 patients will take about 2 years. Considering that the survival of these patients is rather short, median of 2 years for glioma 3-4, complete follow-up will be available for the majority of the highest glioma stages, those who are most likely to develop leukoencephalopathy.

The study will be mainly observational with a follow-up of patients based on classical monitoring. The only additional information collected will come from a CSCT test, a very simple and quick test (90 seconds) to identify mild cognitive dysfunction. A detailed neurological assessment by a neuro-psychologist will be performed before radiotherapy, at 12 and 36 months after radiotherapy and in case of abnormalities of the CSCT.

Methodology

* Study design: Observational prospective cohort of 200 patients, who will be followed every 2-3 months for a period of 3 years after enrolment.
* Eligibility:

Study population: Patients undergoing brain radiotherapy for glioma (stage 3 to 4) between April 2015 and April 2017 at the Mazarin Radiotherapy Department, Pitié-Salpêtrière University Hospital and in the Paul Strauss Institute, Strasbourg .

Before the radiotherapy:

* Description of the cancer: histological type, date of diagnosis, treatment of the cancer: type of surgery (total or partial resection), chemotherapy, etc…
* The radiotherapy planning record: type of radiotherapy (whole brain radiotherapy, stereotactic radiotherapy), total and fractionary delivered doses,
* Results of the CSCT test and of the detailed neuro-psychological tests before treatment Comorbidities will be collected from medical records: hypertension, diabetes, smoking habits, cardiovascular diseases, etc…

After radiotherapy, every 2-3 months:

During routine consultations with neuro-oncologists, the following information will be collected:

* Clinical examination: brain features: intracranial high pressure, progressive focal neurological deficit, epilepsia… and toxicity features: alert symptoms (amnesia, dysexecutive disorders, gait troubles, urinary dysfunction)
* MRI scan of brain: tumor features: progression, stability, response and toxicity features
* Results of the CSCT test

Additional data will be collected:

* Neurocognitive tests results performed during a dedicated consultation with neuropsychologist: before the radiotherapy and 12 and 36 months after the radiotherapy
* Blood samples : before the radiotherapy and 12 and 36 months after the radiotherapy In case of abnormal results at 2 consecutive CSCT tests (-1.5 Standard deviation (SD) of loss) with the exclusion of relapse at MRI, additional cognitive tests will be performed during a dedicated consultation with neuropsychologist. At the end of the follow-up, the vital status of the lost to follow-up patients will be assessed through the National Register for Identification of Physical Persons (RNIPP).

  * Outcomes:

Primary outcome Cognitive dysfunction due to leukoencephalopathy defined by both abnormal results at the CSCT test (confirmed by a complete cognitive test) and a MRI scan of the brain(exclusion of brain tumor relapse).

Secondary outcomes

* Overall death
* Death associated with leukoencephalopathy or cognitive dysfunction ● Data analysis: In this longitudinal study, survival analysis methods will be applied. Occurrence time of the leukoencephalopathy and incidence rates at different follow-up time points (month 6, 12, 18 and 36) will be considered. The Kaplan-Meier estimator will be used to estimate the leukoencephalopathy free survival function. For potential risk factors, hazard ratios associated with outcomes will be estimated using Cox models.

Specificity and sensitivity of the CSCT will be assessed in comparison with complete cognitive test (gold standard)

This project will involve the Neurology department and in the Radiotherapy department in the Pitié Salpétrière University Hospital and in the Paul Strauss Institute

ELIGIBILITY:
Inclusion Criteria:

* - diagnosis of glioma (stage 3 to 4)
* both genders
* age > 18 years
* treatment by radiotherapy and chemotherapy
* clinical monitoring post radiotherapy in Neurology Department, Pitié-Salpêtrière University Hospital and in the radiotherapy department of the Paul Strauss Institute.

Exclusion Criteria:

* - other neurological tumors and brain metastases
* psychiatric severe illness, including severe depression

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult patients treated by radiotherapy and chemotherapy for a glioma stade IV in the Hospital Pitié Salpetreière or in the Paul Strauss hospital from April 2015 to April 2017 will be included.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2015-04; Primary Completion 2018-04 (Estimated); Study Completion 2020-04 (Estimated)

PRIMARY OUTCOMES:
decrease of 1.5 SD of Compurerized Speed Cognitive test | before radiotherapy, at 12 and 36 months

SECONDARY OUTCOMES:
sensitivity and specificity of the Compurerized Speed Cognitive test | at the inclusion time (before radiotherapy), at 12 and 36 months
  comparison of the CSCT result with the results of the complete neurocognitive evaluation.
dosimetric prognostic factors of neurocognitive defects | at the inclusion time (before radiotherapy), and at 12 and 36 months
  collection of histograms of dose-volumes of specific organs and areas based on data from radiotherapy treatment plan.
levels of biomarkers before and after radiotherapy | at the inclusion time (before radiotherapy), , at 12 and 36 months
  levels of homocysteine, protein S100B,specific isoprostanes (8,12-iso-iPF2α-VI),micro RNA, microparticules
radiological prognostic factors of neurocognitive defects | at the inclusion time (before radiotherapy), and at 12 and 36 months
  white matter abnormalities and cortical atrophy.The white matter lesion quantification will follow the procedure described by Wahlund et al (Wahlund 2001) using a 4 points scale (0: no lesion; 1: focal lesions; 2: beginning confluence of lesion; 3: diffuse involvement of the entire region). The cortical atrophy quantification will follow the procedure described by Pasquier et al (Pasquier 1996) using a 4 point scale (0: absence of atrophy; 1: mild atrophy; 2: moderate atrophy; 3: severe atrophy).

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Hopital Pitié Salpétriere, Paris
  - Centre paul Strauss, Strasbourg

REFERENCES:
- [Derived] Durand T, Jacob S, Lebouil L, Douzane H, Lestaevel P, Rahimian A, Psimaras D, Feuvret L, Leclercq D, Brochet B, Tamarat R, Milliat F, Benderitter M, Vayatis N, Noel G, Hoang-Xuan K, Delattre JY, Ricard D, Bernier MO. EpiBrainRad: an epidemiologic study of the neurotoxicity induced by radiotherapy in high grade glioma patients. BMC Neurol. 2015 Dec 18;15:261. doi: 10.1186/s12883-015-0519-6. PMID 26684198